CLINICAL TRIAL: NCT03110562
Title: A Phase 3 Randomized, Controlled, Open-label Study of Selinexor, Bortezomib, and Dexamethasone (SVd) Versus Bortezomib and Dexamethasone (Vd) in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: Bortezomib, Selinexor, and Dexamethasone in Patients With Multiple Myeloma
Acronym: BOSTON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-023
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory Multiple Myeloma; RRMM; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — selinexor; Bortezomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Primary part is parallel (SVd vs Vd treatment arm). Participants who received Vd were allowed to cross-over to receive either SVd or SdX treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SVd Arm: Selinexor + Bortezomib + Dexamethasone (Experimental): Participants received a fixed oral dose of 100 milligrams (mg) selinexor tablets (5 tablets of 20 mg each) once weekly (QW) on Days 1, 8, 15, 22, and 29 of each 35-day cycle, along with subcutaneous (SC) injection of 1.3 milligrams per square meter (mg/m^2) bortezomib QW on Days 1, 8, 15, and 22 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone twice weekly (BIW) on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
  Interventions: Drug: Selinexor; Drug: Bortezomib; Drug: Dexamethasone
- Vd Arm: Bortezomib + Dexamethasone (Experimental): Participants received SC injection of 1.3 mg/m^2 bortezomib on Days 1, 4, 8, and 11 of each 21-day cycle for the first 8 cycles, followed by greater than or equal to (>=) 9 cycles on Days 1, 8, 15, and 22 of each 35-day cycle, and received oral dose of 20 mg dexamethasone BIW on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for the first 8 cycles and for cycles >= 9 on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone
- SVdX Arm: Selinexor + Bortezomib + Dexamethasone (Experimental): Participants in the VD arm who had IRC-confirmed PD and were able to tolerate continued bortezomib treatment had crossed over to receive fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle, along with SC injection of 1.3 mg/m^2 bortezomib QW on Days 1, 8, 15, and 22 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
  Interventions: Drug: Selinexor; Drug: Bortezomib; Drug: Dexamethasone
- SdX Arm: Selinexor + Dexamethasone (Experimental): Participants in the VD arm who had IRC-confirmed PD and were unable to tolerate continued bortezomib treatment had crossed over to receive fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
  Interventions: Drug: Selinexor; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — oral 100 mg dose
  Arms: SVd Arm: Selinexor + Bortezomib + Dexamethasone; SVdX Arm: Selinexor + Bortezomib + Dexamethasone; SdX Arm: Selinexor + Dexamethasone
Drug: Bortezomib — subcutaneous dose of 1.3 mg/m2
  Other Names: Velcade®
  Arms: SVd Arm: Selinexor + Bortezomib + Dexamethasone; SVdX Arm: Selinexor + Bortezomib + Dexamethasone; Vd Arm: Bortezomib + Dexamethasone
Drug: Dexamethasone — oral dose of 20mg

SUMMARY:
This Phase 3, 2-arm, randomized, active comparator-controlled, open-label, multicenter study will compare the efficacy and health-related quality of life (HR-QoL) and assess the safety of selinexor plus bortezomib (Velcade) plus low-dose dexamethasone (SVd) versus bortezomib plus low-dose dexamethasone (Vd) in adult patients with RRMM who have received 1 to 3 prior anti-multiple myeloma (MM) regimens. Crossover from the Vd Arm to a treatment that includes selinexor (i.e., SVdX or SdX) will be allowed at the point of IRC-confirmed objective disease progression per the IMWG criteria for patients in the Vd Arm.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed MM with measurable disease per IMWG guidelines as defined by at least 1 of the following:

   1. Serum M-protein ≥ 0.5 g/dL (> 5 g/L) by serum protein electrophoresis (SPEP) or for immunoglobulin (Ig) A myeloma, by quantitative serum IgA levels; or
   2. Urinary M-protein excretion at least 200 mg/24 hours; or
   3. Serum free light chain (FLC) ≥ 100 mg/L, provided that the serum FLC ratio is abnormal (normal FLC ratio: 0.26 to 1.65).
2. Had at least 1 prior anti-MM regimen and no more than 3 prior anti-MM regimens. Induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 anti-MM regimen.
3. Documented evidence of progressive MM (based on the Investigator's determination according to the modified IMWG response criteria) on or after their most recent regimen.
4. Prior treatment with bortezomib or other Proteasome Inhibitor (PI) is allowed, provided all of the following criteria are met:

   1. Best response achieved with prior bortezomib at any time was ≥ PR and with the last PI (PI therapy (alone or in combination) was ≥ PR, AND
   2. Participant did not discontinue bortezomib due to ≥ Grade 3 related toxicity, AND
   3. Must have had at least a 6-month PI-treatment-free interval prior to Cycle 1 Day 1 (C1D1) of study treatment.
5. Must have an ECOG Status score of 0, 1, or 2.
6. Written informed consent in accordance with federal, local, and institutional guidelines.
7. Age ≥18 years.
8. Resolution of any clinically significant non-hematological toxicities (if any) from previous treatments to ≤ Grade 1 by C1D1. Patients with chronic, stable Grade 2 non-hematological toxicities may be included following approval from the Medical Monitor.
9. Adequate hepatic function within 28 days prior to C1D1.

   1. Total bilirubin <1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of <3 × ULN), and
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to <2 × ULN.
10. Adequate renal function within 28 days prior to C1D1 (estimated creatinine clearance [CrCl] of ≥20 mL/min, calculated using the formula of Cockroft and Gault):

(140-Age) × Mass (kg)/(72 × creatinine mg/dL) Multiply by 0.85 if the patient is female, or if CrCl is ≥20 mL/min as measured by 24-hour urine collection.

11. Adequate hematopoietic function within 7 days prior to C1D1: total white blood cell (WBC) count ≥1500/mm3, absolute neutrophil count ≥1000/mm3, hemoglobin ≥8.5 g/dL and platelet count ≥75,000/mm3 (patients for whom < 50% of bone marrow nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of bone marrow nucleated cells are plasma cells).

1. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.
2. Patients must have:

   * At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and
   * At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment.

However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.

12. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

1. Prior exposure to a SINE compound (i.e. an XPO-1 inhibitor), including selinexor.
2. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) during the 5 years prior to randomization. Cancer treated with curative intent for >5 years previously and without evidence of recurrence will be allowed.
3. Has any concurrent medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
4. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to C1D1. Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
5. Active plasma cell leukemia.
6. Documented systemic light chain amyloidosis.
7. MM involving the central nervous system.
8. Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome.
9. Spinal cord compression.
10. Greater than Grade 2 neuropathy or ≥ Grade 2 neuropathy with pain at baseline, regardless of whether or not the patient is currently receiving medication
11. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
12. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy (including investigational therapies) ≤ 2 weeks prior to C1D1. Localized radiation to a single site at least 1 week before C1D1 is permitted. Glucocorticoids within 2 weeks of C1D1 are permitted. Patients on long-term glucocorticoids during Screening do not require a washout period but must be able to tolerate the specified dexamethasone dose in this study.
13. Prior autologous stem cell transplantation < 1 month or allogeneic stem cell transplantation < 4 months prior to C1D1.
14. Active graft versus host disease (after allogeneic stem cell transplantation) at C1D1.
15. Pregnant or breastfeeding females.
16. Body Surface Area < 1.4 m² at baseline, calculated by the Dubois or Mosteller method.
17. Life expectancy of < 4 months.
18. Major surgery within 4 weeks prior to C1D1.
19. Active, unstable cardiovascular function:

    1. Symptomatic ischemia, or
    2. Uncontrolled clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first-degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
    3. Congestive heart failure of New York Heart Association Class ≥ 3 or known left ventricular ejection fraction < 40%, or
    4. Myocardial infarction within 3 months prior to C1D1.
20. Known active human immunodeficiency virus (HIV) infection or HIV seropositivity
21. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus ribonucleic acid (RNA) or hepatitis B virus surface antigen.
22. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
23. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
24. Contraindication to any of the required concomitant drugs or supportive treatments.
25. Patients unwilling or unable to comply with the protocol, including providing 24-hour urine samples for urine protein electrophoresis at the required time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (157):
- United States (20):
  - Boca Raton Clinical Research (BRCR) Medical Center, Plantation, Florida
  - Emory University, Atlanta, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - McFarland Clinic, Ames, Iowa
  - Stormont Vail Health Care (Cotton O'Neil Cancer Center ), Topeka, Kansas
  - Commonwealth Hematology, Danville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Central Care Cancer Center, Bolivar, Missouri
  - The Valley Hospital Luckow Pavilion, Paramus, New Jersey
  - Mount Sinai, New York, New York
  - The Cancer Institute at St. Francis Hospital, Roslyn, New York
  - Novant-Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - University of Cincinnati Health, Cincinnati, Ohio
  - Southwest Cancer Center of Oklahoma, Lawton, Oklahoma
  - Kaiser Permanente Northwest OR, Portland, Oregon
  - SCOR AnMed Health Cancer Center, Anderson, South Carolina
  - Prairie Lakes Healthcare, Watertown, South Dakota
  - Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
- Australia (8):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Misericordiae Limited and Mater Medical Research, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (5):
  - Medical University Innsbruck, Department of Internal Medicine V (Hematology and Oncology), Innsbruck
  - University Hospital Krems, Department of Internal Medicine II, Krems
  - Medical University of Vienna, Vienna
  - General Hospital Hietzing, Vienna
  - Wilhelminen Hospital, Department of Internal Medicine I, Center for Oncology & Hematology, Vienna
- Belgium (5):
  - Jules Bordet Institute, Brussels
  - UCL Saint-Luc, Brussels
  - University Hospital Ghent, Ghent
  - General Hospital Delta, Roeselare
  - St. Augustinus Hospital, Wilrijk
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment, Sveti Georgi Clinic of Clinical Hematology, Plovdiv
  - University Multiprofile Hospital for Active Treatment, Sveti Ivan Rilski Clinic of Hematology, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases, Clinic of Hematology, Dept. of Clinical Hematology, Sofia
- Canada (11):
  - Tom Baker Cancer Center/ Alberta Health Services, Calgary, Alberta
  - Cross Cancer Institute / University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - North East Cancer Centre Sudbury, Greater Sudbury, Ontario
  - Princess Margaret Cancer Research, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital / McGill University, Montreal, Quebec
  - L'Hôtel-Dieu de Québec, Québec, Quebec
  - Saskatchewan Cancer Agency-Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
- Czechia (6):
  - General University Hospital in Prague, Prague, Prague
  - University Hopsital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Dept. of Hematooncology, Ostrava
  - University Hospital Kralovske Vinohrady, Clinic of Internal Hematology, Prague
- France (8):
  - Hospital Center Departmental La Roche-Sur-Yon, La Roche-sur-Yon
  - Claude Huriez Hospital, Lille
  - South Lyon Hospital Center, Lyon
  - Brabois Adults Hospital, University Hospital Center of Nancy, Nancy
  - Nantes University Hospital Center, Nantes
  - Saint-Louis Hospital, Paris
  - Miletrie Hospital, University Hospital Center of Poitiers, Poitiers
  - Necker Children's Hospital, Department of Adult Hematology, Paris, Île-de-France Region
- Germany (3):
  - University Hospital Freiburg, Department of Internal Medicine I, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Leverkusen gGmbH Medizinisxhe Klinik 3, Leverkusen, North Rhine Westfalia
  - Group Practice for Hematology and Oncology, Dresden, Saxony
- Greece (4):
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - General Hospital of Athens "Evangelismos", Department of Hematology and Lymphoma, Athens
  - University General Hospital of Patra, Pátrai
  - Theageneion Cancer Hospital, Hematology Department, Thessaloniki
- Hungary (5):
  - Semmelweis University, 1st Department of Internal Medicine, Budapest
  - Integrated Szent Istvan and Szent laszlo Hospital, Department of Hematology and Stem Cell Transplantation, Budapest
  - Semmelweis University, 3rd Department of Internal Medicine, Budapest
  - Kaposi Mor Teaching Hospital, 2nd Department of Internal Medicine, Kaposvár
  - Medical Center of the University of Pecs, Department of Hematology, Pécs
- India (20):
  - Regional Cancer Centre, Patna, Bihar
  - Regional Cancer Centre, Thiruvananthapuram, Kerala
  - Prince Aly Khan Hospital, Mumbai, Maharashta
  - Jaslok Hospital and Research Centre, Mumbai, Maharashta
  - Bhaktivedanta Hospital, Thane, Maharashtra
  - IMS & SUM Hospital, Bhubaneswar, Odisha
  - Postgraduate Institute of Medical Education & Research (PGIMER), Chandigarh, Punjab
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Cancer Institute, Chennai, Tamil Nadu
  - SRM Institute of Medical Sciences, Chennai, Tamil Nadu
  - Saveetha Medical College Hospital, Chennai, Tamil Nadu
  - G. Kuppuswamy Naidu Hospital, Coimbatore, Tamil Nadu
  - Asviratham Speciality Hospital, Madurai, Tamil Nadu
  - Meenakshi Mission Hospital, Madurai, Tamil Nadu
  - Yashoda Hospital, Hyderabad, Telangana
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata, West Bengal
  - Nil Ratan Sircar (NRS) Medical College, Kolkata, West Bengal
  - TATA Memorial Centre, Kolkata, West Bengal
  - Rajiv Gandhi Cancer Hospital, New Delhi
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (9):
  - Hospital Santa Maria of Terni, Terni, Umbria
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Polyclinic S. Orsola-Malpighi, Department of Hematology, Oncology and Laboratory Medicine, Operative Unit of Hematology - Cavo, Bologna
  - University Hospital Careggi, Department of Hematology, Florence
  - University Hospital San Martino, IRCCA, Dept. of Integrative Cancer Therapies, Operative Unit of Clinical Hematology, Genoa
  - Hospital Niguerda Ca Granda, Department of Hematology and Oncology, Hematology Unit, Milan
  - Umberto I Polyclinic of Rome, Department of Cellular Biotechnology and Hematology, Hematology Center, Rome
  - University Hospital San Giovanni Battista of Turin, Turin
- Poland (7):
  - Jan Biziel University Hospital #2 in Bydgoszcz, Department of Hematology, Bydgoszcz
  - Independent Public Healthcare Facility Municipal Hospital Group in Chorzow, Department of Hematology, Chorzów
  - University Hospital in Krakow, Teaching Unit of the Hematology Department, Krakow
  - Nicolaus Copernicus Memorial Provincial Specialist Hospital in Lodz, Department of Hematology, Lodz
  - Independent Public Teaching Hospital No.1 in Lublin, Department of Hematology-Oncology and Bone Marrow Transplantation, Lublin
  - St. John of Dukla Oncology Center of Lublin, Department of Hematology, Lublin
  - Military Institute of Medicine, Department of Internal Medicine and Hematology, Warsaw
- Romania (3):
  - Hyperclnical MedLife PDR Vulturului Brasov, Hematology Department, Brasov
  - Colentina Clinical Hospital, Department of Hematology, Bucharest
  - Bucharest University Emergency Hospital, Department of Hematology, Bucharest
- Russia (4):
  - S.P. Botkin City Clinical Hospital, Moscow
  - N.A. Semashko Central Clinical Hospital #2 under OJSC Russian Railways, Moscow
  - First I.P. Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - V.A. Almazov North-West Federal Medical Research Center, Chemotherapy of Oncohematology Diseases and Bone Marrow Transplantation Department #1, Saint Petersburg
- Serbia (5):
  - Clinical Center of Serbia, Clinic of Hematology, Belgrade
  - Institute of Oncology and Radiology of Serbia, Clinic of Medical Oncology, Belgrade
  - Clinical Center Kragujevac, Clinic of Hematology, Kragujevac
  - Clinical Center Nis, Clinic of Hematology and Clinical Immunology, Niš
  - Clinical Center of Vojvodina, Clinic of Hematology, Novi Sad
- Spain (6):
  - University Hospital of the Canary Islands, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Catalan Institute of Oncology (ICO) Badalona, Badalona
  - University Hospital of Vall d'Hebron, Barcelona
  - University Hospital Infanta Leonor, Department of Hematology, Madrid
  - University Clinical Hospital of Salamanca, Department of Hematology, Salamanca
  - University Hospital Virgen del Rocio (HUVR), Seville
- Ukraine (7):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostic Hematology Center, Department of Hematology, Cherkasy
  - City Clinical Hospital No.4 of Dnipro City Council, City hematology center, Dnipropetrovsk
  - BMT Kiev Center, Kiev
  - Kiev Cancer Institute, Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Department of Hematology with Laboratory Group, Lviv
  - Vinnytsia M.I. Pyrohov Regional Clinical Hospital, Department of Hematology, Vinnytsia
  - O.F. Herbachevskyi Regional Clinical Hospital, Hematology Department with Intensive Therapy Wards, Zhytomyr
- United Kingdom (14):
  - Belfast Heatlh & Social Care Trust Belfast City Hospital, Belfast, Northern Ireland
  - NHS Tayside Ninewells Hospital, Dundee, Scotland
  - Cardiff & Vale University Health Board University Hospital of Wales, Cardiff, Wales
  - University Hospitals Birmingham NHS Foundation Trust Queen Elizabeth Hospital, Birmingham
  - The Leeds Teaching Hospitals NHS Trust St. James University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust Royal Leicester Infirmary, Leicester
  - Royal Liverpool & Broadgreen University Hospital NHS Trust Royal Liverpool University Hospital, Liverpool
  - London North West Healthcare NHS Trust Northwick Park Hospital, London
  - University College London, London
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - The Royal Wolverhampton NHS Trust New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jagannath S, Delimpasi S, Grosicki S, Van Domelen DR, Bentur OS, Spicka I, Dimopoulos MA. Association of Selinexor Dose Reductions With Clinical Outcomes in the BOSTON Study. Clin Lymphoma Myeloma Leuk. 2023 Dec;23(12):917-923.e3. doi: 10.1016/j.clml.2023.08.018. Epub 2023 Aug 29. PMID 37743180
- [Derived] Schiller GJ, Lipe BC, Bahlis NJ, Tuchman SA, Bensinger WI, Sutherland HJ, Lentzsch S, Baljevic M, White D, Kotb R, Chen CI, Rossi A, Biran N, LeBlanc R, Grosicki S, Martelli M, Gunsilius E, Spicka I, Stevens DA, Facon T, Mesa MG, Zhang C, Van Domelen DR, Bentur OS, Gasparetto C. Selinexor-Based Triplet Regimens in Patients With Multiple Myeloma Previously Treated With Anti-CD38 Monoclonal Antibodies. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):e286-e296.e4. doi: 10.1016/j.clml.2023.06.001. Epub 2023 Jun 5. PMID 37393120
- [Derived] Delimpasi S, Mateos MV, Auner HW, Gavriatopoulou M, Dimopoulos MA, Quach H, Pylypenko H, Hajek R, Leleu X, Dolai TK, Sinha DK, Venner CP, Benjamin R, Garg MK, Doronin V, Levy Y, Moreau P, Chai Y, Arazy M, Shah J, Shacham S, Kauffman MG, Richardson PG, Grosicki S. Efficacy and tolerability of once-weekly selinexor, bortezomib, and dexamethasone in comparison with standard twice-weekly bortezomib and dexamethasone in previously treated multiple myeloma with renal impairment: Subgroup analysis from the BOSTON study. Am J Hematol. 2022 Mar 1;97(3):E83-E86. doi: 10.1002/ajh.26434. Epub 2021 Dec 29. No abstract available. PMID 34882831
- [Derived] Richard S, Chari A, Delimpasi S, Simonova M, Spicka I, Pour L, Kriachok I, Dimopoulos MA, Pylypenko H, Auner HW, Leleu X, Usenko G, Hajek R, Benjamin R, Dolai TK, Sinha DK, Venner CP, Garg M, Stevens DA, Quach H, Jagannath S, Moreau P, Levy M, Badros A, Anderson LD Jr, Bahlis NJ, Facon T, Mateos MV, Cavo M, Chang H, Landesman Y, Chai Y, Arazy M, Shah J, Shacham S, Kauffman MG, Grosicki S, Richardson PG. Selinexor, bortezomib, and dexamethasone versus bortezomib and dexamethasone in previously treated multiple myeloma: Outcomes by cytogenetic risk. Am J Hematol. 2021 Sep 1;96(9):1120-1130. doi: 10.1002/ajh.26261. Epub 2021 Jul 5. PMID 34062004
- [Derived] Mateos MV, Gavriatopoulou M, Facon T, Auner HW, Leleu X, Hajek R, Dimopoulos MA, Delimpasi S, Simonova M, Spicka I, Pour L, Kriachok I, Pylypenko H, Doronin V, Usenko G, Benjamin R, Dolai TK, Sinha DK, Venner CP, Garg M, Stevens DA, Quach H, Jagannath S, Moreau P, Levy M, Badros AZ, Anderson LD Jr, Bahlis NJ, Cavo M, Chai Y, Jeha J, Arazy M, Shah J, Shacham S, Kauffman MG, Richardson PG, Grosicki S. Effect of prior treatments on selinexor, bortezomib, and dexamethasone in previously treated multiple myeloma. J Hematol Oncol. 2021 Apr 13;14(1):59. doi: 10.1186/s13045-021-01071-9. PMID 33849608
- [Derived] Auner HW, Gavriatopoulou M, Delimpasi S, Simonova M, Spicka I, Pour L, Dimopoulos MA, Kriachok I, Pylypenko H, Leleu X, Doronin V, Usenko G, Hajek R, Benjamin R, Dolai TK, Sinha DK, Venner CP, Garg M, Stevens DA, Quach H, Jagannath S, Moreau P, Levy M, Badros A, Anderson LD Jr, Bahlis NJ, Facon T, Mateos MV, Cavo M, Chai Y, Arazy M, Shah J, Shacham S, Kauffman MG, Richardson PG, Grosicki S. Effect of age and frailty on the efficacy and tolerability of once-weekly selinexor, bortezomib, and dexamethasone in previously treated multiple myeloma. Am J Hematol. 2021 Jun 1;96(6):708-718. doi: 10.1002/ajh.26172. Epub 2021 May 3. PMID 33755235
- [Derived] Grosicki S, Simonova M, Spicka I, Pour L, Kriachok I, Gavriatopoulou M, Pylypenko H, Auner HW, Leleu X, Doronin V, Usenko G, Bahlis NJ, Hajek R, Benjamin R, Dolai TK, Sinha DK, Venner CP, Garg M, Gironella M, Jurczyszyn A, Robak P, Galli M, Wallington-Beddoe C, Radinoff A, Salogub G, Stevens DA, Basu S, Liberati AM, Quach H, Goranova-Marinova VS, Bila J, Katodritou E, Oliynyk H, Korenkova S, Kumar J, Jagannath S, Moreau P, Levy M, White D, Gatt ME, Facon T, Mateos MV, Cavo M, Reece D, Anderson LD Jr, Saint-Martin JR, Jeha J, Joshi AA, Chai Y, Li L, Peddagali V, Arazy M, Shah J, Shacham S, Kauffman MG, Dimopoulos MA, Richardson PG, Delimpasi S. Once-per-week selinexor, bortezomib, and dexamethasone versus twice-per-week bortezomib and dexamethasone in patients with multiple myeloma (BOSTON): a randomised, open-label, phase 3 trial. Lancet. 2020 Nov 14;396(10262):1563-1573. doi: 10.1016/S0140-6736(20)32292-3. PMID 33189178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 165 investigative sites in 21 countries. A total of 402 participants were enrolled and randomized, of which 399 participants received SVd treatment (195 participants) or Vd treatment (204 participants).
Pre-assignment Details: Following confirmation of progressive disease (PD) by the Independent Review Committee (IRC), 204 participants in the safety population who received Vd treatment were allowed to cross over to receive either SVdX treatment (66 participants) or SdX treatment (14 participants).
Groups:
- SdX Arm: Selinexor + Dexamethasone: Participants in the VD arm who had IRC-confirmed PD and were unable to tolerate continued bortezomib treatment had crossed over to receive fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
Period: Initial Treatment Period
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone | SVdX Arm: Selinexor + Bortezomib + Dexamethasone | SdX Arm: Selinexor + Dexamethasone
Started | 195 | 207 | 0 | 0
Treated | 195 | 204 | 0 | 0
Intent-to-treat (ITT) Population (The ITT population consisted of all participants who were randomized to the study treatment, regardless of whether or not they received the study treatment.) | 195 | 207 | 0 | 0
Safety Population (The safety population consisted of all participants who had received at least 1 dose of the study treatment.) | 195 | 204 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 195 | 207 | 0 | 0
Not completed — Disease Progression | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 39 | 41 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 74 | 82 | 0 | 0
Not completed — Lost to Follow-up | 13 | 8 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0
Not completed — Participants withdrawn due to company goals | 59 | 67 | 0 | 0
Not completed — Other | 5 | 4 | 0 | 0
Not completed — Randomized but never treated | 0 | 3 | 0 | 0
Period: Crossover Period
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone | SVdX Arm: Selinexor + Bortezomib + Dexamethasone | SdX Arm: Selinexor + Dexamethasone
Started | 0 | 0 | 66 (66 participants in the safety population who crossed over from the Vd arm to the SVdX treatment arm.) | 14 (14 participants in the safety population who crossed over from the Vd arm to the SdX treatment arm.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 66 | 14
Not completed — Disease Progression | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 6
Not completed — Death | 0 | 0 | 37 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 1
Not completed — Participants withdrawn due to company goals | 0 | 0 | 19 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all participants who were randomized to the study treatment, regardless of whether or not they received the study treatment.
Groups:
- SVd Arm: Selinexor + Bortezomib + Dexamethasone: Participants received a fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle, along with SC injection of 1.3 mg/m^2 bortezomib QW on Days 1, 8, 15, and 22 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
- Vd Arm: Bortezomib + Dexamethasone: Participants received SC injection of 1.3 mg/m^2 bortezomib on Days 1, 4, 8, and 11 of each 21-day cycle for the first 8 cycles, followed by >= 9 cycles on Days 1, 8, 15, and 22 of each 35-day cycle, and received oral dose of 20 mg dexamethasone BIW on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for the first 8 cycles and for cycles >= 9 on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
- Total: Total of all reporting groups
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone | Total
Number analyzed (Participants) | 195 | 207 | 402
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.56) | 66.7 (9.35) | 66.0 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 92 | 172
  Male | 115 | 115 | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 25 | 25 | 50
  Race: Black or African American | 4 | 7 | 11
  Race: White | 161 | 165 | 326
  Race: Other | 0 | 1 | 1
  Race: Missing | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 6 | 5 | 11
  Ethnicity: Not Hispanic or Latino | 171 | 188 | 359
  Ethnicity: Not Reported | 14 | 11 | 25
  Ethnicity: Unknown | 4 | 2 | 6
  Ethnicity: Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: SVd/Vd Arm: Progression-free Survival (PFS) as Assessed by Independent Review Committee (IRC)
Description: PFS was defined as time from date of randomization until the first date of IRC-confirmed PD, per International Myeloma Working Group (IMWG) response criteria, or death due to any cause, whichever occurs first. PD included increase of 25% from lowest confirmed response value in 1 or more of the following criteria: a) serum M-protein with absolute increase of >= 0.5 gram per deciliter (g/dL); b) serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; c) urine M-protein (absolute increase must be >= 200 mg per 24 hours); d) in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be greater than [>] 10 mg/dL); e) in participants without measurable serum and urine M-protein levels and without measurable involved FLC levels: bone marrow plasma cell percentage irrespective of baseline status (absolute increase must be >=10%).
Time Frame: From date of randomization until IRC-confirmed documented PD or death, censored date, whichever occurred first (up to 33 months)
Population: ITT population consisted of all participants who were randomized to the study treatment, regardless of whether or not they received the study treatment. Data was not planned to be reported for SVdx arm and Sdx arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Months | 13.93 [11.73 to NA] — Upper limit of 95% CI was not estimable due to low number of events. | 9.46 [8.11 to 10.78]
Statistical Analysis 1: Comparison: SVd Arm: Selinexor + Bortezomib + Dexamethasone vs Vd Arm: Bortezomib + Dexamethasone; Test type: Superiority; p = 0.0075, Stratified Log-rank Test — One Sided P-value; Stratified for prior PI therapies, number of prior of anti-MM regimens and R-ISS Stage at screening; Hazard Ratio (HR) = 0.7020, 95% CI 2-sided [0.5279 to 0.9335] — Based on stratified Cox Proportional Hazard model with Efron's Method of handling ties

2. Secondary Outcome: SVd/Vd Arm: Overall Response Rate (ORR) as Assessed by IRC
Description: ORR was defined as the percentage of the participants who achieved any confirmed partial response (PR) or better PR, complete response (CR), very good partial response (VGPR) or stringent complete response (sCR) based on the IRC's response outcome assessments, according to the International Myeloma Working Group (IMWG) response criteria, before IRC-confirmed PD or initiating a new MM treatment. PR: >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; or stringent complete response (sCR): CR as defined as Normal free light chain (FLC) ratio + Absence of clonal cells by immunohistochemistry.
Time Frame: From date of randomization until disease progression or initiating a new MM treatment (up to 33 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Percentage of participants | 76.4 [69.8 to 82.2] | 62.3 [55.3 to 68.9]
Statistical Analysis 1: Comparison: SVd Arm: Selinexor + Bortezomib + Dexamethasone vs Vd Arm: Bortezomib + Dexamethasone; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — One Sided P-value; Analysis using Cochran-Mantel-Haenszel test stratified by region, prior PI therapies, number of prior anti-MM regimens, and R-ISS stage at screening; Odds Ratio (OR) = 1.9626, 95% CI 2-sided [1.2641 to 3.0471]

3. Secondary Outcome: SVd/Vd Arm: Percentage of Participants With Response Rate of Very Good Partial Response (VGPR) or Better Based on IRC Assessment
Description: Response rate was defined as percentage of participants with responses of VGPR, at any time prior to IRC-confirmed PD or initiating a new MM treatment. VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: From date of randomization until confirmed PD or initiating a new MM treatment (up to 33 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Percentage of participants | 44.6 [37.5 to 51.9] | 32.4 [26.0 to 39.2]
Statistical Analysis 1: Comparison: SVd Arm: Selinexor + Bortezomib + Dexamethasone vs Vd Arm: Bortezomib + Dexamethasone; Test type: Superiority; p = 0.0082, Cochran-Mantel-Haenszel — One Sided P-value; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.6594, 95% CI 2-sided [1.0993 to 2.5049]

4. Secondary Outcome: SVd/Vd Arm: Number of Participants With at Least One Grade Greater Than or Equal to [>=] 2 Peripheral Neuropathy Events
Description: Peripheral neuropathy events was assessed using the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. The grade ranges from Grade 1 (mild, asymptomatic, or mild symptoms) to Grade 5 (death related to an adverse event). Grade 2 indicates a moderate condition that may require minimal intervention and can limit certain daily activities. Grade 3 represents severe symptoms that are not immediately life-threatening but may lead to hospitalization and restrict self-care activities. Grade 4 denotes life-threatening consequences requiring urgent intervention. Number of participants experiencing at least one Grade >= 2 peripheral neuropathy event have been reported.
Time Frame: From first dose of study treatment to 30 days after the last dose of study treatment inclusive, or the day before the start of new anti-MM treatment, whichever occurs first (up to 33 months)
Population: Safety population included of all participants who had received at least 1 dose of the study treatment. Data was not planned to be reported for SVdx arm and Sdx arm.
Measure: Count of Participants; unit: Participants
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 204
Participants | 41 | 70
Statistical Analysis 1: Comparison: SVd Arm: Selinexor + Bortezomib + Dexamethasone vs Vd Arm: Bortezomib + Dexamethasone; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — One Sided P-value; Odds Ratio (OR) = 0.5042, 95% CI 2-sided [0.3216 to 0.7906] — Stratified by Prior PI therapies (Yes or No), Number of prior anti-MM regimens (1 or >1), and R-ISS stage at study entry (R-ISS Stage III versus R-ISS Stage I or II)

5. Secondary Outcome: SVd/Vd Arm: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until either the date of death due to any cause or until the participant is lost to follow-up, for all participants.
Time Frame: From date of randomization to the date of death or censored date, whichever occurred first (up to 45 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Months | 36.67 [30.19 to NA] — The 95% CI was not available due to insufficient numbers of participants with events. | 32.76 [27.83 to NA] — The 95% CI was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: SVd Arm: Selinexor + Bortezomib + Dexamethasone vs Vd Arm: Bortezomib + Dexamethasone; Test type: Superiority; p = 0.2152, Stratified log-rank test — One Sided P-value; Stratified for prior PI therapies, number of prior anti-MM regimens and R-ISS Stage at screening; Hazard Ratio (HR) = 0.8764, 95% CI 2-sided [0.6313 to 1.2168] — Based on stratified Cox Proportional Hazard model with Efron's Method of handling ties

6. Secondary Outcome: SVd/Vd Arm: Duration of Response (DOR) as Assessed by IRC
Description: DOR was defined as the duration of time from the first occurrence of an IRC confirmed response of at least (>=) PR until the first date of IRC-confirmed PD or death due to any cause, whichever occurred first. PR: >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; PD: Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >= 5 g/dL; Urine M-protein (absolute increase must be >= 200 mg per 24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: From the first documentation of response to the first documentation of PD or death, whichever occurred first (up to 45 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Months | 17.28 [12.55 to 26.25] | 12.88 [9.26 to 15.77]

7. Secondary Outcome: SVdX Arm: Overall Response Rate (ORR1) as Assessed by IRC During SVdX Treatment
Description: ORR was defined as the percentage of the participants who achieved a confirmed partial response or better (i.e., PR, VGPR, CR, or sCR) based on the IRC's response outcome assessments, according to the IMWG response criteria. PR: >=50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >=90% or <200 mg per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow; or sCR: CR as defined as Normal FLC ratio+ Absence of clonal cells in bone marrow biopsy by immunohistochemistry.
Time Frame: From date of first SVdX treatment until disease progression or initiating a new MM treatment (up to 33 months)
Population: The SVdX population consisted of a subset of participants in the Vd arm of the safety population who crossed over from the Vd arm to SVdX treatment after IRC confirmation of PD on Vd and had received at least 1 dose of selinexor. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SVdX Arm: Selinexor + Bortezomib + Dexamethasone
Number analyzed (Participants) | 63
Percentage of participants | 19.0 [10.2 to 30.9]

8. Secondary Outcome: SVdX Arm: Progression Free Survival1 (PFS1) as Assessed by IRC During SVdX Treatment
Description: PFS1 is defined as the duration of time from the date of the first dose of the SVd treatment after crossover from the Vd arm until the first date of PD or death due to any cause, whichever occurred first. PD included increase of 25% from lowest confirmed response value in 1 or more of the following criteria: a) serum M-protein with absolute increase of >= 0.5 gram per deciliter (g/dL); b) serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; c) urine M-protein (absolute increase must be >= 200 mg per 24 hours); d) in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be greater than [>] 10 mg/dL); e) in participants without measurable serum and urine M-protein levels and without measurable involved FLC levels: bone marrow plasma cell percentage irrespective of baseline status (absolute increase must be >=10%).
Time Frame: From date of first SVdX treatment until IRC-confirmed documented PD or death or censored date, whichever occurred first (up to 33 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVdX Arm: Selinexor + Bortezomib + Dexamethasone
Number analyzed (Participants) | 63
Months | 3.91 [3.48 to 6.93]

9. Secondary Outcome: SVd/Vd Arm: Time-to-next-treatment (TTNT) in Participants Randomized to the SVd and Vd Arm Who Received Treatment After SVd/Vd
Description: TTNT is defined as the duration from date of randomization to start of next anti-MM treatment or death, whichever occurs first. For patients without an event, their follow-up time will be censored at the date of discontinuation from study, or last participating visit on or before database cutoff date, whichever occurs first.
Time Frame: From date of randomization to start of next anti-MM treatment or death, whichever occurred first (up to 33 months)
Population: The ITT population consisted of all participants who were randomized to the study treatment, regardless of whether or not they received the study treatment. Data was not planned to be reported for SVdx arm and Sdx arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 195 | 207
Months | 16.13 [13.93 to NA] — The 95% CI was not available due to insufficient numbers of participants with events. | 10.84 [9.82 to 13.40]

10. Secondary Outcome: SVd/Vd Arm: Time To Response (TTR) in Participants Randomized to the SVd and Vd Arm
Description: TTR was defined as duration from randomization to the date of first IRC-confirmed PR or better (i.e., PR, VGPR, CR, or sCR) before IRC-confirmed PD or initiating a new MM treatment per IMWG response criteria. The participants who do not achieve IRC-confirmed PR or better response will be censored at the date of last disease assessment on or before database cutoff date. PR: >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; or sCR: Normal free light chain (FLC) ratio + Absence of clonal cells by immunohistochemistry.
Time Frame: From randomization to the date of first IRC-confirmed PR or better (i.e., PR, VGPR, CR, or sCR), whichever occurred first (up to 33 months)
Population: The ITT population consisted of all patients who were randomized to the study treatment, regardless of whether or not they received the study treatment. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Data was not planned to be reported for SVdx arm and Sdx arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 149 | 129
Months | 1.41 [1.35 to 1.51] | 1.61 [1.51 to 2.14]

11. Secondary Outcome: SVd/Vd/SVdx Arm: Progression Free Survival 2 (PFS 2) in Participants Randomized to the SVd and Vd Arm Who Received Post-SVd/Vd/SVdX Treatment
Description: PFS 2 was defined as the duration of time from the date of the first dose of the treatment after SVd/Vd/SVdX until the first date of PD on treatment after SVd/Vd/SVdX or death due to any cause, whichever occurred first. PD included increase of 25% from lowest confirmed response value in 1 or more of the following criteria: a) serum M-protein with absolute increase of >= 0.5 gram per deciliter (g/dL); b) serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; c) urine M-protein (absolute increase must be >= 200 mg per 24 hours); d) in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be greater than [>] 10 mg/dL); e) in participants without measurable serum and urine M-protein levels and without measurable involved FLC levels: bone marrow plasma cell percentage irrespective of baseline status (absolute increase must be >=10%).
Time Frame: From date of first dose of post-SVd/Vd/SVdX treatment to the date of first PD on post-SVd/Vd/SVdX treatment, or death due to any cause (up to 33 months)
Population: The ITT population consisted of all patients who were randomized to the study treatment, regardless of whether or not they received the study treatment. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Data was not planned to be reported for Sdx arm.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Vd Arm (Non-Crossover): Bortezomib + Dexamethasone: Participants who did not cross over were included and received SC injection of 1.3 mg/m^2 bortezomib on Days 1, 4, 8, and 11 of each 21-day cycle for the first 8 cycles, followed by >= 9 cycles on Days 1, 8, 15, and 22 of each 35-day cycle, and received oral dose of 20 mg dexamethasone BIW on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for the first 8 cycles and for cycles >= 9 on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm (Non-Crossover): Bortezomib + Dexamethasone | SVdX Arm: Selinexor + Bortezomib + Dexamethasone
Number analyzed (Participants) | 69 | 42 | 31
Months | 6.60 [5.39 to 9.43] | 8.84 [5.78 to NA] — The 95% CI was not available due to insufficient numbers of participants with events. | 3.88 [2.79 to NA] — The 95% CI was not available due to insufficient numbers of participants with events.

12. Secondary Outcome: SVd/Vd Arm: Change From Baseline in Participant-Reported Peripheral Neuropathy (PN) Assessed by European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire- Chemotherapy-Induced PN 20 (EORTC- QLQ-CIPN20) Total Scores
Description: The EORTC QLQ-CIPN20 instrument is a 20-item QoL instrument, which has been developed to elicit patients' experience of symptoms and functional limitations related to CIPN. The QLQ-CIPN20 contains 20 items assessing sensory (9 items), motor (8 items), and autonomic symptoms (3 items) containing a 4-point Likert scale (1= not at all, 2= a little, 3= quite a bit, and 4= very much), participants indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. Sensory raw scale scores range from 1 to 36, motor raw scale scores range from 1 to 32, and autonomic raw scale scores range from 1 to 12 for men and 1-8 for women (erectile function item is excluded). All scale scores are linearly converted to a total score with range of 0-100 scale, with higher scores indicating more symptom burden.
Time Frame: Svd Arm: Baseline up to End of treatment (EOT) (at Day 820); Vd Arm: Baseline up to EOT (at Day 848)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone
Number analyzed (Participants) | 71 | 58
Score on a Scale
  Total Sensory Score: Change at EOT | 3.38 (12.436) | 11.17 (19.069)
  Total Motor Score: Change at EOT | 3.56 (14.513) | 9.02 (18.662)
  Total Autonomic Score: Change at EOT: number analyzed (Participants) | 71 | 57
  Total Autonomic Score: Change at EOT | 10.41 (22.201) | 10.92 (25.306)

ADVERSE EVENTS:
Time Frame: From date of randomization up to 45 months
Description: In other adverse events section, System Organ Classes for SVD and VD arms were recorded as per MedDRA version 24.1 and remaining events were recorded as per MedDRA version 22.0.
Groups:
- SVd Arm: Selinexor + Bortezomib + Dexamethasone: Participants received a fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle, along with SC injection of 1.3 mg/m^2 bortezomib QW on Days 1, 8, 15, and 22 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death or sponsor decision to terminate the study.
- SdX Arm: Selinexor + Dexamethasone: Participants in the VD arm who had IRC-confirmed PD and were unable to tolerate continued bortezomib treatment had crossed over to receive fixed oral dose of 100 mg selinexor tablets (5 tablets of 20 mg each) QW on Days 1, 8, 15, 22, and 29 of each 35-day cycle, along with SC injection of 1.3 mg/m^2 bortezomib QW on Days 1, 8, 15, and 22 of each 35-day cycle, and an oral dose of 20 mg of dexamethasone BIW on Days 1, 2, 8, 9, 15, 16, 22, 23, 29, and 30 of each 35-day cycle until PD confirmed by the IRC, investigator or participant decision to discontinue study treatment, pregnancy, unacceptable AEs or toxicity that could not be managed by supportive care, withdrawal of consent, death, or sponsor decision to terminate the study.
Arm/Group | SVd Arm: Selinexor + Bortezomib + Dexamethasone | Vd Arm: Bortezomib + Dexamethasone | SVdX Arm: Selinexor + Bortezomib + Dexamethasone | SdX Arm: Selinexor + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 74/195 | 82/204 | 37/66 | 3/14
Serious Adverse Events (participants affected / at risk) | 109/195 | 79/204 | 28/66 | 7/14
Other Adverse Events (participants affected / at risk) | 193/195 | 197/204 | 65/66 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SVd Arm: Selinexor + Bortezomib + Dexamethasone (N=195) | Vd Arm: Bortezomib + Dexamethasone (N=204) | SVdX Arm: Selinexor + Bortezomib + Dexamethasone (N=66) | SdX Arm: Selinexor + Dexamethasone (N=14)
Anaemia (Blood and lymphatic system disorders) | 7 | 3 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 9 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 0
General physical health deterioration (General disorders) | 3 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 24 | 25 | 4 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 3 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 1 | 0
Septic shock (Infections and infestations) | 4 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 2 | 1
Respiratory syncytial virus infection (Infections and infestations) | 2 | 1 | 1 | 1
Urosepsis (Infections and infestations) | 3 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 2 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Vascular dementia (Nervous system disorders) | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0
Reactive psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SVd Arm: Selinexor + Bortezomib + Dexamethasone (N=195) | Vd Arm: Bortezomib + Dexamethasone (N=204) | SVdX Arm: Selinexor + Bortezomib + Dexamethasone (N=66) | SdX Arm: Selinexor + Dexamethasone (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 120 | 56 | 33 | 4
Anaemia (Blood and lymphatic system disorders) | 72 | 45 | 30 | 3
Neutropenia (Blood and lymphatic system disorders) | 30 | 12 | 14 | 1
Leukopenia (Blood and lymphatic system disorders) | 11 | 3 | 4 | 0
Tachycardia (Cardiac disorders) | 10 | 3 | 0 | 0
Cataract (Eye disorders) | 43 | 16 | 14 | 2
Vision blurred (Eye disorders) | 13 | 9 | 0 | 0
Visual impairment (Eye disorders) | 14 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 98 | 21 | 26 | 4
Diarrhoea (Gastrointestinal disorders) | 63 | 53 | 19 | 3
Constipation (Gastrointestinal disorders) | 33 | 35 | 7 | 3
Vomiting (Gastrointestinal disorders) | 39 | 10 | 16 | 2
Abdominal pain (Gastrointestinal disorders) | 15 | 12 | 3 | 1
Fatigue (General disorders) | 82 | 37 | 15 | 3
Asthenia (General disorders) | 48 | 25 | 10 | 0
Oedema peripheral (General disorders) | 23 | 29 | 5 | 2
Pyrexia (General disorders) | 29 | 25 | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 38 | 29 | 8 | 1
Bronchitis (Infections and infestations) | 22 | 19 | 4 | 0
Nasopharyngitis (Infections and infestations) | 23 | 11 | 2 | 1
Pneumonia (Infections and infestations) | 16 | 12 | 5 | 2
Urinary tract infection (Infections and infestations) | 13 | 9 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 12 | 9 | 3 | 1
Weight decreased (Investigations) | 51 | 25 | 18 | 6
Alanine aminotransferase increased (Investigations) | 13 | 7 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 70 | 10 | 19 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 10 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 13 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 7 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 6 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 28 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 17 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 20 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 12 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 66 | 99 | 16 | 2
Dizziness (Nervous system disorders) | 24 | 10 | 4 | 0
Headache (Nervous system disorders) | 20 | 13 | 0 | 2
Paraesthesia (Nervous system disorders) | 5 | 15 | 1 | 2
Insomnia (Psychiatric disorders) | 31 | 32 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 31 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 1 | 1
Hypertension (Vascular disorders) | 17 | 16 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 13 | 4 | 4 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 6 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 11 | 7 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 6 | 0 | 0
Dysgeusia (Nervous system disorders) | 13 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 16 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 0 | 0
Hypotension (Vascular disorders) | 10 | 12 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03110562/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT03110562/SAP_001.pdf